CLINICAL TRIAL: NCT01297036
Title: Open Label, Randomized, Single-dose, Crossover Study to Evaluate the Pharmacokinetic Characteristics of Donepezil Between Two Donepezil Products, Aricept® Tablet and Neuropezil ODT, in Healthy Subjects
Brief Title: Pharmacokinetic Comparisons of Two Donepezil Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Chong Kun Dang Pharmaceutical Corp. (Industry)
Responsible Party: Ji-Young Park, MD/Associate Professor of Clinical Pharmacology, Anam Hospital, Dept. of Clincial Pharmacology, Anam Hospital, Korea University College of Medicine, Seoul, Korea
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 121HPS07D_03
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2008-01

CONDITIONS: Alzheimer Disease
Keywords: Pharmacokinetics; Bioequivalence; Donepezil
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil; Long-Term Synaptic Depression; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reference arm (Active Comparator): Treated with Reference (Aricept, 10 mg donepezil tablet)
  Interventions: Drug: Donepezil, 10 mg tablet
- Test arm (Experimental): Treated with Test (Neuropezil, 10 donepezil ODT, orally disintegrating tablet)
  Interventions: Drug: Donepezil, ODT 10 mg

INTERVENTIONS:
Drug: Donepezil, ODT 10 mg — Test- Donepezil Hydrochloride 10 mg Tablet single dose
  Other Names: Neuropezil ODS; developed by Chong Kun Dang Co, Ltd.
  Arms: Test arm
Drug: Donepezil, 10 mg tablet — Reference: Donepezil Hydrochloride 10 mg Tablet
  Other Names: Aricept:; Manufactured by Dae Woong harm. Co. Ltd, Seoul, Korea
  Arms: Reference arm

SUMMARY:
To compare the relative bioavailability and pharmacokinetic characteristics of a newly developed donepezil formulation with a conventional formulation in healthy subjects with a single dose, randomized, open-label, 2-sequence -2period crossover study.

DETAILED DESCRIPTION:
This single dose, open label, balanced, randomized, two-treatment, two-period, two-sequence, crossover study was conducted to compare the relative bioavailability and pharmacokinetic characteristics of a newly developed formulation with a conventional formulation in healthy subjects.

For this, a single-center, randomized, single-dose, open-label, 2-way crossover study with a 21-day washout period was conducted in 22 healthy volunteers. Plasma samples for the analysis of donepezil were collected up to 240 h after drug administration. Participants received either reference or test drug formulation of 10 mg donepezil in the first period and the alternative formulation in the second period. Plasma concentrations of donepezil were determined by validated high-performance liquid chromatography coupled to tandem mass spectrometry detection. Pharmacokinetic parameters, including Cmax and AUC, were determined by noncompartmental analysis. Analysis of variance (ANOVA) was carried out using log-transformed Cmax and AUC, and the mean ratios and their 90% confidence intervals (CI) were calculated. According to regulatory requirements set forth by Korea and the US Food and Drug Administration, products meet the criteria for bioequivalence if the 90% CIs of the mean ratios for Cmax and AUC are within the range of 0.80 to 1.25.

ELIGIBILITY:
Inclusion Criteria:

* Males age 20 to 45 years
* Body weight > 45 kg with +/- 20% of ideal body weight
* Signed and dated informed consent form which meets all criteria of current FDA and KFDA regulations

Exclusion Criteria:

* subjects with acute conditions.
* presence of history affecting ADME
* Clinically significant history or current evidence of a hepatic, renal, gastrointestinal, or hematologic abnormality
* Hepatitis B, hepatitis C, or HIV infection revealed on the laboratory findings
* Any other acute or chronic disease
* A history of hypersensitivity to donepezil
* A history of alcohol or drug abuse
* Participation in another clinical trial within 3 months
* smoked >10 cigarettes daily
* consumption over 5 glasses daily of beverages containing xanthine derivatives
* use of any medication having the potential to affect the study results within 10 days before the start of the study.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2008-01; Primary Completion 2008-03 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
donepezil pharmacokinetics: peak plasma concentrations (Cmax) | 240 hours
donepezil pharmacokinetics: Area under the time vs. plasma concentration curve from 0 to 240 hr(AUCall) | 240 hours
donepezil pharmacokinetics: Area under the time vs. plasma concentration curve from 0 to infinity(AUCinf) | 240 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Young Park, MD, PhD, Principal Investigator — Anam Hospital, Korea Univeristy College of Medicine
Locations (1):
- Dept. of Clinical Pharmacology & Toxicology, Anam Hospital, Korea University College of Medicine, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Kim KA, Lim JL, Kim C, Park JY. Pharmacokinetic comparison of orally disintegrating and conventional donepezil formulations in healthy Korean male subjects: a single-dose, randomized, open-label, 2-sequence, 2-period crossover study. Clin Ther. 2011 Jul;33(7):965-72. doi: 10.1016/j.clinthera.2011.06.003. Epub 2011 Jul 2. PMID 21723605